CLINICAL TRIAL: NCT00254176
Title: Effect of Cysteine Supplementation on Glutathione Production in Critically Ill Neonates
Brief Title: Cysteine Supplementation in Critically Ill Neonates
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Stephen B. Shew, M.D., UCLA School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-12-035-05; 5K08HD052885-04 (NIH)
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Sepsis; Bronchopulmonary Dysplasia; Necrotizing Enterocolitis; Retinopathy of Prematurity; Systemic Inflammatory Response Syndrome
Keywords: Neonate; Glutathione; Cysteine; Sepsis; Stable Isotope
MeSH Terms: conditions — Sepsis; Bronchopulmonary Dysplasia; Enterocolitis, Necrotizing; Retinopathy of Prematurity; Systemic Inflammatory Response Syndrome | interventions — amino-acid, glucose, and electrolyte solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cysteine (Active Comparator): Subjects that receive cysteine
  Interventions: Dietary Supplement: Parenteral cysteine-HCl supplementation
- No-cysteine placebo (Placebo Comparator): Subjects that do not receive cysteine but an isonitrogenous placebo
  Interventions: Dietary Supplement: Placebo - added premasol

INTERVENTIONS:
Dietary Supplement: Parenteral cysteine-HCl supplementation — cysteine-HCl supplementation 121 mg per kg per day
  Arms: Cysteine
Dietary Supplement: Placebo - added premasol — Premasol 121 mg per kg per day
  Other Names: Trophamine
  Arms: No-cysteine placebo

SUMMARY:
Critically ill babies less than 1 month of age have deficient amounts of the antioxidant glutathione and a high incidence of disease associated with oxidative injury compared to healthy babies. These diseases include but are not limited to damage to the eyes, lungs, and intestines. Frequently becoming chronic and potentially life threatening, these diseases result in a significantly decreased quality of life to the infant along with increased costs to the infant's family and society.

The amino acid cysteine comprises a third of the tripeptide glutathione and directly influences glutathione production. Older children ill with infection and stable, premature neonates administered cysteine supplementation to their diet have been previously shown to increase their glutathione production and concentrations. Furthermore, cysteine supplementation in the ill children resulted in a quicker resolution of their illness.

Although most critically ill babies require IV nutrition (i.e., TPN) before and during their illness, commercially available TPN does not include cysteine as a significant nutrient. Cysteine has effectively become a safe and standard supplement to routine TPN in a few major hospitals in the U.S.

The purpose of this study is to evaluate the ability of cysteine supplementation to increase glutathione production and concentrations in critically ill babies. Furthermore, the investigators want to evaluate whether cysteine supplementation results in less oxidative tissue injury and ultimately less severe illnesses. The study will enroll babies admitted to the UCLA Medical Center Neonatal Intensive Care Unit (NICU) and they will be chosen at random and in a blinded fashion to receive either cysteine or non-cysteine supplementation to their routine TPN. Small blood samples along with a single 6 hour infusion of a non-radioactive, stable isotope labeled amino acid will be used to measure the production of glutathione as well as other compounds in the blood to give a quantitative assessment to the severity of illness. Clinical information relevant to the babies' illness and subsequent recovery will be recorded.

The results will be compared between cysteine vs. non-cysteine groups and before vs. after individual supplementation. By demonstrating the effect of cysteine supplementation on glutathione production, the incidence and/or severity of disease from oxidative injury in critically ill babies may be decreased if glutathione production is improved.

DETAILED DESCRIPTION:
Specific Aims:

Critically ill neonates have demonstrated low concentrations of the antioxidant glutathione and a high incidence of disease associated with oxidative injury compared to healthy neonates. Cysteine is considered to be a conditionally essential amino acid for neonates and is the rate limiting substrate for the synthesis of glutathione. We hypothesize that parenterally-fed, critically ill neonates administered cysteine supplementation will have higher concentrations of total glutathione, lower ratios of oxidized to reduced glutathione, higher glutathione synthetic rates, lower levels of inflammatory cytokine production and lipid peroxidation, and decreased severity of disease associated with oxidative injury compared to similarly ill parenterally fed neonates without cysteine supplementation. To test this hypothesis, critically ill, parenterally fed neonates assigned randomly to receive a cysteine or an isonitrogenous cysteine-free supplement to their TPN (total parenteral nutrition) regimen will be prospectively studied in a double-blind fashion according to the following specific aims:

1. to measure total concentrations of erythrocyte glutathione, oxidized to reduced (GSSG:GSH) erythrocyte glutathione ratios, and the in vivo fractional and absolute synthetic rates of erythrocyte glutathione utilizing a [13C]-glycine tracer,
2. to measure plasma interleukin-6 (IL-6), tumor necrosis factor (TNF-a), and malondialdehyde concentrations as determinants of illness severity and degree of oxidative injury reflected by lipid peroxidation,
3. and, to measure duration of mechanical ventilation, duration of supplemental oxygen, and duration of hospitalization as the primary clinical outcomes of disease severity.

By demonstrating whether cysteine supplementation increases the synthesis and concentration of glutathione along with the subsequent decrease in oxidative injury and associated disease, the widespread morbidity and mortality for vulnerable, critically ill neonates may be improved.

Background:

Critically ill neonates treated in the Neonatal Intensive Care Unit (NICU), whether premature or full term, experience a high incidence of diseases that may be secondary to or exacerbated by oxidative injury. These include a variety of multi-factorial disease processes such as respiratory distress syndrome (RDS), persistent pulmonary hypertension (PPHN), chronic lung disease (CLD), sepsis, meconium aspiration, retinopathy of prematurity (ROP), and necrotizing enterocolitis (NEC). Within NICUs across the U.S. per year, Neonatologists and Pediatric Surgeons care for an estimated 100,000 critically ill neonates, of which approximately 35% are full-term and up to 20% will ultimately expire of their illnesses despite major advances in neonatal care. Some neonatal diseases are well known to have a varying prevalence according to neonatal maturity. Premature neonates more commonly suffer from RDS, CLD, ROP and NEC, with the most susceptible being the extremely premature. However, 10-15% of neonates who develop NEC are full-term and have a resultant mortality rate of up to 35%. Furthermore, other disease processes causing significant respiratory distress (e.g., PPHN, pneumonia, and meconium aspiration) more commonly occur in full-term neonates.

The high morbidity of these diseases has a significant impact for the neonate, their parents, and society in general. Neonatal survivors of critical illness who are without obvious neurologic injury have been found later to have lower IQ's, increased behavioral problems, decreased ability to perform normal activities of daily living, decreased scholastic abilities, and decreased health-related quality of life compared to healthy children. The economic burden to the parents and society from the care of these neonatal illnesses can be astounding. For example, the economic costs of neonatal healthcare alone can increase 32-71% when a critically ill neonate has NEC compared to appropriately matched controls without NEC. Adjusted for inflation to the year 2005, an additional expense of approximately $281,666 is expected for every NEC survivor prior to discharge from the NICU (equivalent to $8.45 million per year for a single large healthcare center). Similarly, the continued healthcare costs of critically ill neonates even after discharge can be insurmountable. Children who were survivors of a critical illness as a premature neonate have been shown to require increased utilization of Pediatric Intensive Care Unit (PICU) resources (e.g., mechanical ventilation), increased length of ICU care, and more frequent readmission to the PICU compared to other PICU patients.

Although cysteine is a non-essential amino acid made from methionine via cystathionine in children and adults, most premature and term neonates have a decreased capacity to synthesize cysteine due to their low expression of the rate limiting enzyme cystathionase. As a result, plasma cysteine and cystine concentrations in critically ill neonates are low compared to healthy infants. Unfortunately, plasma cysteine concentrations of neonates receiving cysteine-free TPN remain low despite generous methionine intakes and relatively high plasma methionine concentrations in TPN fed neonates. This is particularly relevant since cysteine is the limiting substrate for the synthesis of the principal intracellular antioxidant in the body - glutathione.

Intracellular glutathione serves many roles in the cell including protection against oxidative damage caused by free radicals through glutathione peroxidase and detoxification of electrophilic metabolites through multiple glutathione transferases. Thereby, the level of glutathione in a specific organ or tissue is thought to be a major determinant of the vulnerability of that organ or tissue to oxidative stress. Although the majority of whole body glutathione is produced in hepatocytes, most cells, including the erythrocyte, have the equivalent capacity to synthesize glutathione de novo from the 3 amino acids cysteine, glutamate, and glycine utilizing (-glutamylcysteine and glutathione synthetases. The active form of glutathione (reduced or GSH) is also regenerated from recycling of oxidized glutathione (glutathione disulfide or GSSG) through glutathione reductase. However, when the use of reduced glutathione exceeds the capacity of regeneration, the GSSG is expelled from the cell and intracellular glutathione stores are depleted.

Regardless of the degree of stress or neonatal weight, critically ill neonates have activity levels of these glutathione synthetic enzymes comparable to those of adults. Furthermore, these neonates demonstrate unimpeded ability to transport amino acids, including cysteine derivatives, across cellular membranes. Hence, neonates demonstrate the capacity to synthesize glutathione given the appropriate substrates are available. Despite the potential ability to synthesize glutathione, low glutathione concentrations and high ratios of GSSG:GSH have been demonstrated from the blood, lung, and intestine of critically ill neonates in multiple studies. Consequently, a likely limiting factor in the production of glutathione for critically ill neonates is the availability of cysteine in their diet.

Most critically ill neonates receive their nutrition solely through the parenteral route during the acute duration of their illness, from a few days to weeks of post-natal life. Unfortunately, there is no parenteral amino acid formulation commercially available in the U.S. which includes cysteine as a significant nutrient. This is because cysteine is relatively unstable and cystine (i.e., cysteine dimer) is insoluble in aqueous solution. However, cysteine supplementation to TPN is possible in the form of cysteine-HCl if given within 24 hours prior to infusion. Subsequent provision of cysteine in this manner results in higher plasma cysteine concentrations in critically ill neonates. Although cysteine-HCl supplementation to TPN has been shown to be possible and safe, it is not routine practice in current neonatal care. Nevertheless, cysteine-HCl supplementation is standard practice in some major neonatal centers in the U.S. in order to augment the calcium and phosphorus solubility in TPN, which further benefits growing infants.

Several in vitro and animal studies demonstrate cysteine supplementation increases glutathione concentrations in the blood, liver, and intestines. Cysteine supplementation to premature neonatal erythrocytes in cell cultures have demonstrated increased glutathione concentrations compared to non-cysteine supplemented controls. Malloy et. al. have shown cysteine-HCl supplemented TPN-fed beagle pups have higher concentrations of plasma cysteine and hepatic glutathione than unsupplemented TPN-fed pups. Similarly, Pollack et. al. have demonstrated intestinal glutathione concentrations significantly increase in premature newborn rabbits administered cysteine-HCl supplementation compared to non-supplemented controls. Moreover, the colonic glutathione concentrations were found to be similar to those of maternally reared, term newborn rabbits.

As a clinical corollary, human studies in stressed adults with acute respiratory distress syndrome have demonstrated elevated concentrations of glutathione and improvements in recovery after cysteine supplementation. Septic and malnourished children supplemented with enteral cysteine have demonstrated increased glutathione concentrations and in vivo glutathione synthetic rates measured utilizing a novel non-radioactive, stable isotope methodology. Furthermore, the septic children supplemented with cysteine resolved their illnesses quicker than their unsupplemented counterparts. These studies suggest that cysteine-HCl supplementation may improve glutathione production and decrease oxidative stress in critically ill neonates.

There has yet to be an investigation confirming that improved glutathione concentrations and in vivo glutathione synthetic rates occur in critically ill neonates supplemented with cysteine-HCl and that these perturbations lead to a decrease in the amount of oxidative tissue injury that these patients endure. This gap in studies serves as a perfect setting for our proposed randomized, blinded, placebo-controlled trial that is adequately powered to detect a pre-determined difference between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated neonates of all gestational ages and birth weights
* less than 1 month of postnatal age admitted to the NICU
* SNAP (Score of Neonatal Acute Physiology) > 10
* projected requirement for continued parenteral nutrition of at least 1 week duration

Exclusion Criteria:

* renal or hepatic failure
* requiring insulin administration
* requiring extracorporeal life support
* known inherited metabolic disorders
* known uniformly fatal congenital anomalies

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2006-09; Primary Completion 2011-03 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Total RBC glutathione | 0 days, 7 days, 60 days

SECONDARY OUTCOMES:
Tumor necrosis factor (TNF) | 0 days, 7 days, 60 days
Interleukin-6 (IL-6) | 0 days, 7 days, 60 days
Oxygen dependency | through to discharge
Ventilation dependency | through to discharge
Erythrocyte oxidized:reduced glutathione ratio | 0 days, 7 days, 60 days
In vivo erythrocyte glutathione synthetic rate | 7 days, 60 days
Plasma malondialdehyde concentration | 0 days, 7days, 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Shew, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Medical Center, Mattel Childrens Hospital, Los Angeles, California, United States

REFERENCES:
- [Background] Miller RG, Keshen TH, Jahoor F, Shew SB, Jaksic T. Compartmentation of endogenously synthesized amino acids in neonates. J Surg Res. 1996 Jun;63(1):199-203. doi: 10.1006/jsre.1996.0247. PMID 8661197
- [Background] Shew SB, Keshen TH, Jahoor F, Jaksic T. Assessment of cysteine synthesis in very low-birth weight neonates using a [13C6]glucose tracer. J Pediatr Surg. 2005 Jan;40(1):52-6. doi: 10.1016/j.jpedsurg.2004.09.011. PMID 15868558
- [Background] Badaloo A, Reid M, Forrester T, Heird WC, Jahoor F. Cysteine supplementation improves the erythrocyte glutathione synthesis rate in children with severe edematous malnutrition. Am J Clin Nutr. 2002 Sep;76(3):646-52. doi: 10.1093/ajcn/76.3.646. PMID 12198013
- [Background] Miller RG, Jahoor F, Jaksic T. Decreased cysteine and proline synthesis in parenterally fed, premature infants. J Pediatr Surg. 1995 Jul;30(7):953-7; discussion 957-8. doi: 10.1016/0022-3468(95)90320-8. PMID 7472952
- [Background] Lyons J, Rauh-Pfeiffer A, Ming-Yu Y, Lu XM, Zurakowski D, Curley M, Collier S, Duggan C, Nurko S, Thompson J, Ajami A, Borgonha S, Young VR, Castillo L. Cysteine metabolism and whole blood glutathione synthesis in septic pediatric patients. Crit Care Med. 2001 Apr;29(4):870-7. doi: 10.1097/00003246-200104000-00036. PMID 11373484
- [Background] Zlotkin SH, Anderson GH. The development of cystathionase activity during the first year of life. Pediatr Res. 1982 Jan;16(1):65-8. doi: 10.1203/00006450-198201001-00013. PMID 7070878
- [Background] Pollack PF, Rivera A Jr, Rassin DK, Nishioka K. Cysteine supplementation increases glutathione, but not polyamine, concentrations of the small intestine and colon of parenterally fed newborn rabbits. J Pediatr Gastroenterol Nutr. 1996 May;22(4):364-72. doi: 10.1097/00005176-199605000-00005. PMID 8732899
- [Background] Moison RM, Haasnoot AA, van Zoeren-Grobben D, Berger HM. Red blood cell glutathione and plasma sulfhydryls in chronic lung disease of the newborn. Acta Paediatr. 1997 Dec;86(12):1363-9. doi: 10.1111/j.1651-2227.1997.tb14914.x. PMID 9475317
- [Background] Vina J, Vento M, Garcia-Sala F, Puertes IR, Gasco E, Sastre J, Asensi M, Pallardo FV. L-cysteine and glutathione metabolism are impaired in premature infants due to cystathionase deficiency. Am J Clin Nutr. 1995 May;61(5):1067-9. doi: 10.1093/ajcn/61.4.1067. PMID 7733030
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765